CLINICAL TRIAL: NCT02614053
Title: Continuous Non Invasive Monitoring of Both Plethysmography Variability Index and Total Hemoglobin During Cesarean Section for Antepartum Hemorrhage As a Method For Early Detection of Bleeding
Brief Title: Plethysmography Variability Index Monitoring for Parturients With Antepartum Hemorrhage
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, ahmed elsakka, lecturer of anaesthesia faculty of medicine cairo university, Kasr El Aini Hospital
Other Study IDs: mp3
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Antepartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Masimo Radical-7™ Pulse CO-Oximeter — a device collecting data regarding PVI, PI & spHB

SUMMARY:
The purpose of this study is to evaluate the use of continuous noninvasive intraoperative plethesmography variability index in conjunction with Hemoglobin levels monitoring using Masimo Radical-7™ Pulse CO-Oximeter during elective cesarean sections in patients with antepartum and intrapartum hemorrhage as a guide for fluid and blood transfusion practice .

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologist (ASA) Physical status I - II.
* patients aged from 18 to 40 years
* full-term multigravida parturients
* antepartum hemorrhage
* singleton fetus

Exclusion Criteria:

* Patients with known cardiac problem
* peripheral circulatory failure of the upper extremities
* significant liver disease
* significant renal disease
* significant coagulopathy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: parturients with antepartum hemorrhage admitted for cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Pleth Variability Index | 8 months

SECONDARY OUTCOMES:
hemoglobin level | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: nadia yo helmy, md, Study Director — professor of anaesthesia cairo university